CLINICAL TRIAL: NCT04882462
Title: A Multicenter, Single-arm Study of Sintilimab and Nimotuzumab Combined With Chemotherapy for the Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Sintilimab and Nimotuzumab Combined With Chemotherapy for the Treatment of R/M HNSCC.
Acronym: Carpp-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other); Cinda Biopharmaceutical (Suzhou) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-IST-H&N-20210318
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — nimotuzumab; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: Nimotuzumab; Drug: Sintilimab; Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab, 400mg, intravenously every 3 weeks, for at least 18 weeks
Drug: Sintilimab — Sintilimab, 200mg, intravenously every 3 weeks, for at least 18 weeks;
Drug: Chemotherapy drug — Chemotherapy drugs were selected by the investigator, every 3 weeks, for 18 weeks

SUMMARY:
This clinical study is designed as a prospective, open-label, single arm, multicenter study to evaluate the clinical efficacy and safety of Sintilimab and Nimotuzumab in combination with chemotherapy in patients with newly diagnosed recurrent/metastatic head and neck squamous cell carcinoma (R/M HNSCC). The main endpoint is progression free survival (PFS); the secondary endpoint are objective response rate (ORR), disease control rate (DCR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and sign a consent form;
2. Age 18-75 years old, gender unlimited;
3. Histology or imaging diagnosed as R/M HNSCC, patients haven't received any anti-tumor treatment for R/M HNSCC; Including oral cavity cancer, oropharyngeal cancer, hypopharyngeal cancer, laryngeal cancer, nasopharyngeal cancer, paranasal sinus and nasal cavity cancer, etc.;
4. PD-L1 immunohistochemistry and EGFR immunohistochemistry should be performed on tumor tissue samples;
5. according to the efficacy evaluation criteria for solid tumors (RECIST version 1.1), at least one measurable lesion;
6. Not received any previous systemic antitumor therapy for R/M HNSCC. Subjects who had previously received adjuvant/neoadjuvant chemotherapy, or had received radical chemoradiotherapy for advanced disease, were allowed to be enrolled in this study if the interval between disease progression or recurrence and the end of the last treatment (including chemotherapy /EGFR monoclonal antibody /EGFR-TKI/ antiangiogenic agents) was beyond 6 months. Radiotherapy for individual recurrent and/or metastatic lesions cannot be ruled out.
7. ECOG PS 0-2
8. Expected survival time ≥ 3 months;
9. Enough organ function, the participants need to satisfy the following laboratory indicators: 1) nearly 14 days without the use of granulocyte colony stimulating factor, absolute neutrophil count ≥ 1.5 × 109/L; 2) Platelets ≥100×109/L in the case of no blood transfusion in the last 14 days; 3) Hemoglobin ≥9g/dL (90g/L) or≥5.6 mmol/L in the absence of blood transfusion or erythropoietin treatment within the last 14 days; 4) total bilirubin ≤1.5×upper limit of normal (ULN); 5) Aspartate aminotransferase (AST) /alanine aminotransferase (ALT) ≤2.5×ULN, or AST/ALT≤5×ULN in subjects with liver metastasis; 6) Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 mL /min; 7) Good coagulant function; 8) Thyroid function is normal; 9) Myocardial enzyme spectrum is normal;
10. For females of reproductive age, a pregnancy test with negative results should be performed within 3 days prior to receiving the first dosing (cycle 1 day 1);
11. To avoid pregnancy, an effective contraception should used for female patients.

Exclusion Criteria:

1. squamous cell carcinoma of skin;
2. Patients with uncured malignancies other than R/M HNSCC diagnosed within 5 years prior to initial administration;
3. Participating in other clinical studies, or receiving other investigational drugs or using investigational devices within 4 weeks prior to first dosing;
4. Have received any other anti-tumor treatment for R/M HNSCC, including PD-1 inhibitor, PD-L1 inhibitor, CD137 inhibitor, EGFR monoclonal antibody, EGFR-TKI, anti-angiogenic drugs, etc.;
5. Major surgery or chemotherapy was performed within 4 weeks prior to enrollment;
6. Have received immunomodulatory drugs (including thymosin, interferon, interleukin);
7. Active autoimmune disease with systemic therapy (such as glucocorticoids or immunosuppressants) within 2 years prior to initial administration. Alternative therapy (e.g. thyroxine, insulin, etc.) is not considered systemic therapy.
8. Have received systemic glucocorticoid therapy within 7 days prior to enrollment; Note: Physiological dose of glucocorticoids (≤10 mg/ day of prednisone or equivalent drugs) is allowed.
9. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
10. Allergic to the study drugs;
11. Have not fully recovered from toxicity and/or complications caused by any intervention prior to enrollment;
12. History of human immunodeficiency virus (HIV) infection;
13. Untreated active hepatitis B; Note: Hepatitis B patients who meet the following criteria can also be enrolled: 1) HBV DNA<1000 copies /ml (200 IU/ml) prior to enrollment; 2) anti-HBcAg(+), HBsAg (-), anti-HBsAg (-), and HBV DNA(-), prophylactic anti-HBV therapy is not required, but virus reactivation needs to be closely monitored;
14. Active HCV infection;
15. Live vaccine was given within 30 days;
16. Pregnant or lactating women;
17. Any serious or uncontrollable systemic disease;
18. Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 12 months

SECONDARY OUTCOMES:
ORR | Up to 12 months
  objective response rate
DCR | Up to 12 months
  disease control rate
OS | Up to 12 months
  overall survival

OTHER OUTCOMES:
Biomarker | Up to 12 months
  To evaluate the relationship between tumor biomarkers (including but not limited to EGFR or PD-L1 expression, TILs, TMB, HPV status, P16 expression, etc.) and prognosis.